CLINICAL TRIAL: NCT01302158
Title: An Open-label, Randomized Crossover Study to Evaluate the Effect of ASP1941 on the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Glimepiride in Healthy Subjects and Vice Versa
Brief Title: Drug-drug Interaction Study With ASP1941 and Glimepiride
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Disclosure Office Europe, Astellas Pharma Europe BV
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1941-CL-0059; 2009-013172-50 (EudraCT Number)
Record Dates: First submitted 2011-02-21; First posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Healthy Subjects
Keywords: Drug-Drug interaction; ASP1941; Glimepiride; Healthy subjects
MeSH Terms: interventions — ipragliflozin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ASP1941 — oral
Drug: Glimepiride — oral

SUMMARY:
A study to investigate the effect of ASP1941 on the pharmacokinetics and safety of glimepiride (Part A) and to investigate the effect of glimepiride on the pharmacokinetics, safety and pharmacodynamics of ASP1941 (Part B).

DETAILED DESCRIPTION:
Study includes two parts. Part A is to investigate the effect of multiple oral doses of ASP1941 on the pharmacokinetics of glimepiride, and Part B is to investigate the effect of multiple oral doses of glimepiride on the pharmacokinetics of ASP1941.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 and 30 kg/m2, inclusive

Exclusion Criteria:

* Any of the liver function tests above the upper limit of normal
* Pulse <40 or >90 bpm; Systolic Blood Pressure >140 mmHg; Diastolic Blood Pressure > 90 mmHg

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2009-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Effect of multiple doses of ASP1941 on the Pharmacokinetics of glimepiride | 14 days

SECONDARY OUTCOMES:
Effect of multiple doses of glimepiride on the Pharmacokinetics of ASP1941 | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Groningen, Netherlands